CLINICAL TRIAL: NCT04602312
Title: Online RCT Comparing the Effects of Mindfulness, Sham Mindfulness and Book Listening Control on Coronavirus-related Catastrophizing in Adults
Brief Title: How Does Mindfulness Meditation Buffer the Negative Effects of Pain and Suffering in the COVID-19 World? (Healthy Sample)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: University of Sydney (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019000347-S4C
Record Dates: First submitted 2020-10-19; First posted 2020-10-26 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Catastrophizing Coronavirus (COVID-19)
Keywords: Coronavirus-related Catastrophizing
MeSH Terms: conditions — COVID-19 | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: 4 x (2) mixed design, with training (mindfulness vs specific sham mindfulness vs general sham mindfulness vs book listening control, between subjects) and time (pre-treatment vs post-treatment, within-subjects) as factors.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness meditation (Experimental): "focussed attention" mindfulness meditation technique taught as means to reduce coronavirus-related catastrophizing.
  Interventions: Other: Meditation (1 x 20-minute guided audio training)
- Specific sham mindfulness meditation (Sham Comparator): a training session designed to specifically match the real mindfulness training while lacking the proposed active elements of mindfulness training. Delivered as a means to elicit expectancy-mediated (but not mindfulness-mediated) reductions in coronavirus-related catastrophizing.
  Interventions: Other: Meditation (1 x 20-minute guided audio training)
- General sham mindfulness meditation (Sham Comparator): a training session designed to generally match focussed-attention mindfulness meditation while maintaining greater distance from proposed mindfulness mechanisms. Delivered as a means to elicit expectancy-mediated (but not mindfulness-mediated) reductions in coronavirus-related catastrophizing.
  Interventions: Other: Meditation (1 x 20-minute guided audio training)
- Book listening control (No Intervention): this group completes no meditation training. They listen to a spoken excerpt from the audiobook "The Natural History and Antiquities of Selborne"

INTERVENTIONS:
Other: Meditation (1 x 20-minute guided audio training) — Participants will complete a single session of 20-minutes online guided audio-delivered training session of one of the four conditions.
  Arms: General sham mindfulness meditation; Mindfulness meditation; Specific sham mindfulness meditation

SUMMARY:
Both mindfulness meditation and expectancy effects are known to reduce anxiety, stress and catastrophizing, but it is unknown whether and how expectancy effects contribute to the overall effect of mindfulness meditation on these outcomes, especially during significant global events such as the coronavirus pandemic. This study includes four interrelated aims that will probe these effects and interactions.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able to read and understand English

Exclusion Criteria:

* Recurrent pain (two or more days in the last month)
* Chronic pain (pain most days in the last three months)
* Incomplete or invalid data (response time < 32 minutes, failing attention checks)
* Completing the 20-minute training module in < 18 minutes or > 90 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
Coronavirus-related catastrophizing | 40 minutes
  assessed via a covid-19-related catastrophizing scale (CCS; 0=no catastrophizing, 52=highest catastrophizing, 30+=clinically significant catastrophizing)

OTHER OUTCOMES:
Expectancy | 40 minutes
  assessed via self-report questions (0=lowest expectancy, 10=highest expectancy)
Reappraisal | 40 minutes
  assessed via the Cognitive Emotion Regulation Questionnaire (CERQ-R; 4=lowest reappraisal, 20=highest reappraisal)
Mindful observing | 40 minutes
  assessed via the Five Facet Mindfulness Questionnaire Observing subscale (FFMQ-O; 1=lowest observing, 5=highest observing)
Mindful non-reactivity | 40 minutes
  assessed via the Five Facet Mindfulness Questionnaire Non-reacting subscale (FFMQ-NR; 1=lowest non-reactivity, 5=highest non-reactivity)
State Mindfulness | 40 minutes
  assessed via the State Mindfulness Survey (SMS; 1=lowest mindfulness, 21=highest mindfulness)
State Decentering | 40 minutes
  assessed via the Metacognitive Processes of Decentering - State (MpoD-s; 0=lowest decentering, 3=highest decentering)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Day, PhD, Principal Investigator — The University of Queensland
Locations (1):
- Health and Behavioural Sciences, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual trial-related participant data collected during the trial, after de-identification.
Supporting Information: SAP, ICF
Time Frame: Immediately following publication up and for a further 10 years .
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee. Initial contact should be directed to the contact person for scientific enquiries (Mr Jonathan Davies, jonathan.davies@uq.edu.au).
  Note: Requestors will need to sign a data access agreement.
URL: https://sites.google.com/view/uqcovidmeditation

REFERENCES:
- See also: TAKE THE SURVEY NOW - LINK FOR PARTICIPANTS WISHING TO PARTICIPATE — https://sydneypsy.qualtrics.com/jfe/form/SV_6P8sOROQ5eq8SpL?src=CTGC
- See also: INFORMATION ABOUT THE STUDY — https://sites.google.com/view/uqcovidmeditation